CLINICAL TRIAL: NCT01619319
Title: Effects of Cognitive Remediation on Cognition in Young People at Clinical High Risk of Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Jean Addington, M.D., Principal Investigator, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Cognitive Remediation in CHR
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Prodromal Schizophrenia
Keywords: schizophrenia prodrome; clinical high risk of psychosis
MeSH Terms: conditions — Schizotypal Personality Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Remediation Therapy (Experimental): A computerised cognitive remediation intervention called the Brain Fitness program is compared against a placebo intervention consisting of computer games
  Interventions: Other: Cognitive Remediation Therapy
- computer games (Active Comparator): computer games
  Interventions: Other: computer games

INTERVENTIONS:
Other: Cognitive Remediation Therapy — auditory computer games designed to improve the speed at which people react when they hear something and at which they process that information.
  Other Names: Brain Fitness Program
  Arms: Cognitive Remediation Therapy
Other: computer games — computer games that that consist of word puzzles
  Other Names: Hoyle Puzzle and Board Games
  Arms: computer games

SUMMARY:
Onset of psychotic disorders such as schizophrenia, typically occurs during late adolescence or early adulthood often resulting in chronic social and occupational disability. Deficits in cognition and functional outcome often precede the onset of full-blown psychosis although to a lesser degree than observed in schizophrenia. Recent progress in risk identification methodology has enabled reliable detection of persons who appear to be putatively prodromal for psychosis, that is, at clinical high risk (CHR) of developing a psychotic disorder. Since these CHR individuals already evidence cognitive deficits, which increase around the time of conversion, cognition is an excellent treatment target. Furthermore, there is clear evidence, in schizophrenia and in CHR samples, that deficits in cognition are related to poor functional outcome. Thus, treatments targeting cognition may consequently improve functional outcome. The primary aim of the project is to reduce cognitive deterioration and improve cognition among youths at CHR using cognitive remediation and to test the effectiveness of a new cognitive remediation program, the Brain Fitness program, in improving cognition of CHR individuals. A control treatment consisting of video games (VG) will be used. The primary hypothesis is that the BF group will have improved cognition at the end of treatment and 12 months post baseline compared to the VG group. A secondary hypothesis is that improved cognition will be associated with improved functioning. This is a longitudinal, single blind, placebo controlled pilot trial of cognitive remediation in 36 CHR persons. Participants will be randomised to either the BF or VG program, which will be administered over a period of 3 months. Assessments will occur at baseline, post treatment (3 months) and at 12 months after baseline. All subjects will be recruited in year 1 of the project and treatment will be completed by 15 months. The 40 hours of training will occur 4 days a week, for an hour each day, over a period of 10 -12 weeks.

DETAILED DESCRIPTION:
Participants were randomised to either the BFP or a control treatment consisting of commercial computer games (CG). Participants were not blind to group allocation but all cognitive and symptom raters were. The 40 hours of BFP or computer game activity was expected to occur 4 days a week, for an hour each day, over a period of 10-12 weeks. The primary outcome was cognitive function assessed using the MATRICS consensus cognitive battery MCCB) (Nuechterlein and others 2008). The secondary outcome was social and role functioning assessed with Global Functioning: Social and Role scales. All clinical and cognitive assessments using symptom, functioning and cognitive measures were performed at baseline, post-treatment (at 3 months) and at 9-month follow-up (i.e. 9 months post baseline or 6 months after post-treatment assessment).

ELIGIBILITY:
Inclusion Criteria:1.

1. Male or female between 12 and 35 years old.
2. Understand and sign an informed consent (or assent for minors) document in English.
3. Must meet the NAPLS substance use criteria (see guidelines).
4. Meet diagnostic criteria for prodromal syndrome as per COPS Criteria (see below) or if under 19 meet criteria for schizotypal personality disorder.

   -

Exclusion Criteria:

1. Meet criteria for current or lifetime Axis I psychotic disorder, including affective psychoses and psychosis NOS.
2. No current treatment with antipsychotic medication unless it can be clearly demonstrated that the diagnostic prodromal criteria were present prior to the antipsychotic.
3. Impaired intellectual functioning (i.e IQ<70); however those with an IQ in the 65-69 range will be included if the WRAT reading >75.
4. Past or current history of a clinically significant central nervous system disorder that may contribute to prodromal symptoms or confound their assessment.
5. Traumatic Brain Injury that is rated as 7 or above on the Traumatic Brain Injury screening instrument.
6. The diagnostic prodromal symptoms are clearly caused by an Axis 1 disorder, including substance use disorders, in the judgment of the evaluating clinician. Other non-psychotic DSM-IV disorders will not be exclusionary (e.g. substance abuse disorder, major depression, anxiety disorders, Axis II Disorders), as long as the disorder does not account for the diagnosis of prodromal symptoms.

   -

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2010-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) | 12 months
  MATRICS will be used to assess changes in cognition at the end of treatment and 12 months post baseline.

SECONDARY OUTCOMES:
GFS= Global Functioning Scale (GFS): Social and Role | 12 months
  Functioning scales will be used to asses if changes in cognitive function are associated with changes in social and role functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Addington, PhD, Principal Investigator — University of Calgary

REFERENCES:
- See also: Faculty of medicine, University of Calgary — http://www.ucalgary.ca/jaddingt/